CLINICAL TRIAL: NCT04577846
Title: Surgical Site Infection (SSI) Rates in Patients Undergoing Mastectomy Without Reconstruction, a Comparison Among Those Receiving Preoperative Prophylactic Antibiotics Alone Versus Continued Prophylactic Antibiotics Postoperatively-A Multicenter, Double-blinded Randomized Control Trial.
Brief Title: SSI Rates in Patients Undergoing Mastectomy Without Reconstruction- A Multicenter, Double-blinded RCT.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Collaborators: Liaquat National Hospital & Medical College (Other); Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Abida K. Sattar, MD, FACS, Assistant Professor and Section Head, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2020-3627-1407
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Surgical Site Infection
Keywords: mastectomy; antibiotic prophylaxis; surgical site infection; drains
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cephalexin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Active Comparator): The intervention arm will be administered, either Cefazolin iv every 8 hours while NPO or cefalexin 500 mg q8 hours per oral if tolerating a diet.
  Interventions: Drug: Cephalexin 500 MG
- Control (Placebo Comparator): Controls will be provided with initially IV placebo while NPO and then with a placebo capsule filled with inert material for the duration of the drains which usually is about 14 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cephalexin 500 MG — Cefalexin 500 mg PO q8 hours will be continued for the duration of the indwelling drains which usually is about 14 days.
  Arms: Intervention Arm
Drug: Placebo — A placebo capsule filled with inert material for the duration of the drains which usually is about 14 days.
  Arms: Control

SUMMARY:
Breast cancer is the second most prevalent malignancy in the world and an important component of treatment warrants surgical procedures such as mastectomy. Surgical site infections after breast surgery may range from 1-26%, which is high for surgeries that are considered "clean procedures", as defined by the Centers for Disease Control and Prevention (CDC) wound classification system.

Prophylactic antibiotics given before the surgical incision as per Joint Commissions SCIP (Surgical Care Improvement Project) guidelines, have been shown to decrease the rate of postoperative infections in a vast number of patients. There is however, no clear consensus due to lack of evidence on continuation (duration) of prophylactic antibiotics in patients undergoing mastectomy with indwelling drains, and thus antibiotic prescribing practices may vary among breast as well as reconstructive surgeons.

In this trial all patients undergoing mastectomy without immediate reconstruction will receive a single prophylactic dose of preoperative antibiotic, and subsequently, the patients will be randomized to either continue the prophylactic antibiotics or receive a placebo for the duration of indwelling drains. The aim of this trial is to compare the difference in SSI rates between these two study arms as the main outcome. In addition, the factors associated with differing rates of SSI in the intervention and control group will also be identified.

DETAILED DESCRIPTION:
Introduction:

Worldwide, breast cancer comprises 10.4% of all cancer among women, making it the second most common cancer (after lung cancer) and the fifth most common cause of cancer related death. The management of patients as a matter of patient preference or as dictated by extent of disease often warrants a mastectomy.

Reports of surgical site infections after breast surgery including mastectomy may range from 1-26%, which is high for surgeries that are considered "clean procedures". Despite a high rate of surgical site infections, there is no consensus on the continuation/duration of prophylactic antibiotics in patients undergoing mastectomy. Consequently, practices may vary among breast and reconstructive surgeons. Evidence regarding the risk of SSI with the use and duration of indwelling drains is also controversial. The length of prolonged, postoperative antibiotic may also vary by practitioners, some using a pre-defined regimen of about 2-7 days, and others continuing them until the drains are removed.

Most guidelines recommend a single dose of pre-operative antibiotics and continuation after surgery has been discouraged. The use of common or more specific antibiotics for the duration of drains being in place is also controversial. The recommendation by recent national clinical guidelines is to use one dose of pre-procedural antibiotics for mastectomy patients with or without drains. The American Society of Breast Surgeons also does not recommend the continuation of post-surgical antibiotics in the absence of relevant indications. However, practices vary.

Rationale:

Since there is lack of evidence and significant surgeon practice variation despite guidelines developed by leading societies, we propose to study the difference in rates of surgical site infection (SSI) with or without continuation of prolonged post-operative, prophylactic antibiotics in all patients undergoing mastectomy without immediate reconstruction and with indwelling drains.

Aim:

In this trial all patients undergoing mastectomy without immediate reconstruction will receive a single prophylactic dose of preoperative antibiotic, and subsequently, the patients will be randomized to either continue the prophylactic antibiotics or receive a placebo for the duration of indwelling drains. The aim of this trial is to compare the difference in SSI rates between these two study arms as the main outcome. In addition, the factors associated with differing rates of SSI in the intervention and control group will also be identified.

Significance:

Through this study, the investigators will be able to identify the most effective prophylactic regimen to reduce rates of SSI among mastectomy patients with indwelling drains leading to evidence-based and informed decision making.

Primary Objective:

To determine rates of surgical site infection (SSI) in patients in two separate arms of this trial, in which all patients will receive the first prophylactic pre/perioperative antibiotic dose and then be randomized to:

1. Post-operative antibiotic prophylaxis continued for the duration of indwelling drains
2. Those who only receive a single dose of preoperative prophylactic antibiotic.

Secondary Objective:

To identify factors associated with differing rates of SSI in the intervention and control group

Primary Outcome:

Surgical site infection(SSI) rates at the mastectomy wound site or the drain(s) insertion site among patients. In this study SSI will be evaluated using the standard CDC criteria which are as follows:

1. purulent drainage from the incision or drain site;
2. organisms isolated from an aseptically obtained culture of fluid or tissue;
3. deliberate opening of the incision by a surgeon in patients having either tenderness, localized swelling, redness, or warmth; or
4. diagnosis of SSI by the surgeon or study wound assessor (trained research assistant) or
5. prescription of therapeutic antibiotics;
6. Patients clinically diagnosed and documented to have cellulitis.

ELIGIBILITY:
Inclusion Criteria: Patients who will undergo mastectomy (without immediate reconstruction) at AKUH, LNH, and DUHS (with or without axillary surgery), who will have indwelling closed suction drain(s) postoperatively and will give consent to participate in the study

Exclusion Criteria:

* Undergo breast reconstruction
* Who have other medical indications for which they must remain on antibiotics for more than the single preoperative dose
* Those with any history of allergies to beta-lactam drug
* Patients who had an open breast or axillary biopsy/breast conservation in the last 30 days on the ipsilateral side.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Surgical Site Infection (SSI) | up to 30 days.
  Standard CDC criteria:
  1. purulent drainage from the incision or drain site;
  2. organisms isolated from an aseptically obtained culture of fluid or tissue;
  3. deliberate opening of the incision by a surgeon in patients having either tenderness, localized swelling, redness, or warmth; or
  4. diagnosis of SSI by the surgeon or study wound assessor or
  5. prescription of therapeutic antibiotics;
  6. Patients clinically diagnosed and documented to have cellulitis.

OTHER OUTCOMES:
Rates of antibiotic associated side-effects | will be assessed during the follow-up visits between postoperative days 4-8 days for the 1st postoperative visit and subsequently at each routine postoperative visit while the drain is in place, for a maximum of 30 days.
  infections/diarrhea/other side effects

CONTACTS AND LOCATIONS:
Overall Officials: Abida K. Sattar, MD, FACS, Principal Investigator — Aga Khan University
Locations (3):
- Pakistan (3):
  - Dow University of Health Sciences, Karachi, Sindh
  - Aga Khan University Hospital, Karachi, Sindh
  - Liaquat National Hospital, Karachi, Sindh

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared

REFERENCES:
- [Background] Zeeshan S, Ali B, Ahmad K, Chagpar AB, Sattar AK. Clinicopathological Features of Young Versus Older Patients With Breast Cancer at a Single Pakistani Institution and a Comparison With a National US Database. J Glob Oncol. 2019 Mar;5:1-6. doi: 10.1200/JGO.18.00208. PMID 30860954
- [Background] Vilar-Compte D, Jacquemin B, Robles-Vidal C, Volkow P. Surgical site infections in breast surgery: case-control study. World J Surg. 2004 Mar;28(3):242-6. doi: 10.1007/s00268-003-7193-3. Epub 2004 Feb 17. PMID 14961196
- [Background] Throckmorton AD, Boughey JC, Boostrom SY, Holifield AC, Stobbs MM, Hoskin T, Baddour LM, Degnim AC. Postoperative prophylactic antibiotics and surgical site infection rates in breast surgery patients. Ann Surg Oncol. 2009 Sep;16(9):2464-9. doi: 10.1245/s10434-009-0542-1. Epub 2009 Jun 9. PMID 19506959
- [Background] Degnim AC, Scow JS, Hoskin TL, Miller JP, Loprinzi M, Boughey JC, Jakub JW, Throckmorton A, Patel R, Baddour LM. Randomized controlled trial to reduce bacterial colonization of surgical drains after breast and axillary operations. Ann Surg. 2013 Aug;258(2):240-7. doi: 10.1097/SLA.0b013e31828c0b85. PMID 23518704
- [Background] Angarita FA, Acuna SA, Torregrosa L, Tawil M, Escallon J, Ruiz A. Perioperative variables associated with surgical site infection in breast cancer surgery. J Hosp Infect. 2011 Dec;79(4):328-32. doi: 10.1016/j.jhin.2011.08.006. Epub 2011 Nov 3. PMID 22054593
- [Background] Jones DJ, Bunn F, Bell-Syer SV. Prophylactic antibiotics to prevent surgical site infection after breast cancer surgery. Cochrane Database Syst Rev. 2014 Mar 9;(3):CD005360. doi: 10.1002/14651858.CD005360.pub4. PMID 24609957
- [Background] Felippe WA, Werneck GL, Santoro-Lopes G. Surgical site infection among women discharged with a drain in situ after breast cancer surgery. World J Surg. 2007 Dec;31(12):2293-9; discussion 2300-1. doi: 10.1007/s00268-007-9248-3. PMID 17917771
- [Background] Gao YX, Xu L, Ye JM, Wang DM, Zhao JX, Zhang LB, Duan XN, Liu YH. Analysis of risk factors of surgical site infections in breast cancer. Chin Med J (Engl). 2010 Mar 5;123(5):559-62. PMID 20367981
- [Background] Vilar-Compte D, Rosales S, Hernandez-Mello N, Maafs E, Volkow P. Surveillance, control, and prevention of surgical site infections in breast cancer surgery: a 5-year experience. Am J Infect Control. 2009 Oct;37(8):674-9. doi: 10.1016/j.ajic.2009.02.010. Epub 2009 Jun 24. PMID 19556033
- [Background] Teija-Kaisa A, Eija M, Marja S, Outi L. Risk factors for surgical site infection in breast surgery. J Clin Nurs. 2013 Apr;22(7-8):948-57. doi: 10.1111/jocn.12009. Epub 2012 Nov 2. PMID 23121264
- [Background] Thomson DR, Sadideen H, Furniss D. Wound drainage after axillary dissection for carcinoma of the breast. Cochrane Database Syst Rev. 2013 Oct 20;2013(10):CD006823. doi: 10.1002/14651858.CD006823.pub2. PMID 24158902
- [Background] Rotstein C, Ferguson R, Cummings KM, Piedmonte MR, Lucey J, Banish A. Determinants of clean surgical wound infections for breast procedures at an oncology center. Infect Control Hosp Epidemiol. 1992 Apr;13(4):207-14. doi: 10.1086/646511. PMID 1593101
- [Background] Rey JE, Gardner SM, Cushing RD. Determinants of surgical site infection after breast biopsy. Am J Infect Control. 2005 Mar;33(2):126-9. doi: 10.1016/j.ajic.2004.05.004. PMID 15761414
- [Background] Bratzler DW, Dellinger EP, Olsen KM, Perl TM, Auwaerter PG, Bolon MK, Fish DN, Napolitano LM, Sawyer RG, Slain D, Steinberg JP, Weinstein RA; American Society of Health-System Pharmacists (ASHP); Infectious Diseases Society of America (IDSA); Surgical Infection Society (SIS); Society for Healthcare Epidemiology of America (SHEA). Clinical practice guidelines for antimicrobial prophylaxis in surgery. Surg Infect (Larchmt). 2013 Feb;14(1):73-156. doi: 10.1089/sur.2013.9999. Epub 2013 Mar 5. No abstract available. PMID 23461695
- [Background] Hedrick TL, Smith PW, Gazoni LM, Sawyer RG. The appropriate use of antibiotics in surgery: a review of surgical infections. Curr Probl Surg. 2007 Oct;44(10):635-75. doi: 10.1067/j.cpsurg.2007.06.006. No abstract available. PMID 18021817
- [Background] Edwards BL, Stukenborg GJ, Brenin DR, Schroen AT. Use of prophylactic postoperative antibiotics during surgical drain presence following mastectomy. Ann Surg Oncol. 2014 Oct;21(10):3249-55. doi: 10.1245/s10434-014-3960-7. Epub 2014 Aug 20. PMID 25138078
- [Background] Wilcox MH, Mooney L, Bendall R, Settle CD, Fawley WN. A case-control study of community-associated Clostridium difficile infection. J Antimicrob Chemother. 2008 Aug;62(2):388-96. doi: 10.1093/jac/dkn163. Epub 2008 Apr 22. PMID 18434341
- [Background] Wilcox MH, Chalmers JD, Nord CE, Freeman J, Bouza E. Role of cephalosporins in the era of Clostridium difficile infection. J Antimicrob Chemother. 2017 Jan;72(1):1-18. doi: 10.1093/jac/dkw385. Epub 2016 Sep 22. PMID 27659735
- [Background] Thomas C, Stevenson M, Riley TV. Antibiotics and hospital-acquired Clostridium difficile-associated diarrhoea: a systematic review. J Antimicrob Chemother. 2003 Jun;51(6):1339-50. doi: 10.1093/jac/dkg254. Epub 2003 May 13. PMID 12746372
- [Derived] Sattar AK, Zahid N, Shahzad H, Soomro R, Saleem O, Mahmood SF. Impact of duration of antibiotic prophylaxis on rates of surgical site infection (SSI) in patients undergoing mastectomy without immediate reconstruction, comparing a single prophylactic dose versus continued antibiotic prophylaxis postoperatively: a multicentre, double-blinded randomised control trial protocol. BMJ Open. 2021 Jul 9;11(7):e049572. doi: 10.1136/bmjopen-2021-049572. PMID 34244280
- See also: An Updated Meta-Analysis on the Effectiveness of Preoperative Prophylactic Antibiotics in Patients Undergoing Breast Surgical Procedures — https://www.infona.pl/resource/bwmeta1.element.elsevier-c2ba39f4-6e68-34c2-9881-843f77cb211e
- See also: Specifications Manual for Joint Commission National Quality Core Measures — https://www.jointcommission.org/measurement/specification-manuals/
- See also: National Practice Patterns in Preoperative and Postoperative Antibiotic Prophylaxis in Breast Procedures Requiring Drains: Survey of the American Society of Breast Surgeons — http://link.springer.com/article/10.1245/s10434-012-2477-1